CLINICAL TRIAL: NCT00987090
Title: Early-onset and Late-onset Sporadic Alzheimer's Disease (AD) : Variations of the Clinical Profile and Paraclinical Features Depending on the Age at the Onset of Clinical Signs
Brief Title: Early-onset and Late-onset Sporadic Alzheimer's Disease (AD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008/24; 2008-A01213-52
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer's Disease
Keywords: subjects developing symptoms of Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alzheimer Disease (Active Comparator): subjects who have developed symptoms of Alzheimer Disease aged from 45 to 85 years old
  Interventions: Biological: Clinic and neuropsychologic evaluation; Radiation: MRI; Procedure: PET; Biological: Apolipoprotein E genotyping; Biological: Study of cerebrospinal fluid
- Control (Placebo Comparator): subjects without symptoms of Alzheimer Disease aged from 45 to 85 years old.
  Interventions: Biological: Clinic and neuropsychologic evaluation; Radiation: MRI; Procedure: PET; Biological: Apolipoprotein E genotyping

INTERVENTIONS:
Biological: Clinic and neuropsychologic evaluation — evaluation at the inclusion and 18 months after
Radiation: MRI — intervention at the inclusion and 18 months after
Procedure: PET — 18-FDG (18-fluoro-2-deoxyglucose)PET imaging of the brain at the inclusion and 18 months after.
Biological: Apolipoprotein E genotyping — genotyping at the inclusion
Biological: Study of cerebrospinal fluid — intervention at the inclusion
  Arms: Alzheimer Disease

SUMMARY:
Alzheimer's disease (AD) is usually associated with aging, age being the principal identified risk factor. However, younger subjects also develop AD and the prevalence of early onset AD is unknown. It is estimated that about 30 000 subjects develop symptoms of AD before the age of 65 in France. There is evidence that early onset AD differs from AD in older patients. In particular, clinical and neuroimaging studies suggest early involvement of neocortical brain regions and their functions in early onset AD, while mediotemporal areas and memory might be more involved in late onset AD. These differences could partly explain the atypical clinical and imaging features of younger patients, the diagnostic difficulties in these patients and the specific problems related to medical care of this age group. The present study uses a multidisciplinary approach with longitudinal followup in order to establish the impact of age on the clinical and neuroimaging picture of sporadic AD in a multicentric setting. Another aim of the project is to describe for each age group, and in particular for the younger patient group, the functional impact of disability in everyday life on both, patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Arm Alzheimer Disease : first symptoms from 1 to 5 years before the inclusion, Clinical Dementia Rating = 1, efficient contraception for women
* Arm Control : efficient contraception for women

Exclusion Criteria:

* Important general disease : diabetes, neoplasia, alcoholism
* First symptoms less than 1 year or more than 5 years before the inclusion
* Pregnancy, breast feeding

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
to establish the impact of age on the clinical and neuroimaging picture of sporadic Alzheimer Disease in a multicentric setting. | 3 years

SECONDARY OUTCOMES:
to describe for each age group, and in particular for the younger patient group, the functional impact of disability in everyday life on both, patients and caregivers. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: mathieu ceccaldi, Principal Investigator — Assistance Publique - Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France, France